CLINICAL TRIAL: NCT02004561
Title: Outcomes Comparison Between Gastric Band, Laparoscopic Sleeve Gastrectomy, and Gastric Bypass Surgeries in Obese Adolescents
Brief Title: Comparison Between Gastric Band, Laparoscopic Sleeve Gastrectomy, Gastric Bypass Surgeries
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1109009034; 2R01HD028016-20A1 (NIH)
Record Dates: First submitted 2013-11-11; First posted 2013-12-09 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Obese Adolescents
Keywords: bariatric_surgery; pediatric obesity; diabetes
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastric Banding: Patients chose Gastric banding
- Gastric Bypass: Patients chose gastric bypass surgical operation

SUMMARY:
Determine the short and long term safety and efficacy of the Gastric bypass , laparoscopic sleeve gastrectomy, and Gastric banding (LAGB) on severely obese adolescents. The procedure selection is made by the patient or patient and guardian. This is not a randomized trial.

DETAILED DESCRIPTION:
Twenty-six obese adolescents with plans to undergo bariatric surgery for clinical treatment will be recruited for research study during screening process at the Yale Adolescent Bariatric Surgery Clinic. After the appropriate discussion with surgeon, the choice of procedure will be made by subject and legal guardian.

Every bariatric patient must have completed the thorough six-month evaluation period established by the Yale's Adolescent Bariatric Clinic.

This standard of care pre-operative testing provides as a screening tool to ensure every adolescent bariatric patient is mentally and physically appropriate for this surgery.

* Monthly visits with clinician (Pediatric Obesity/Diabetology Expert) and dietician to discuss lifestyle change management and anthropometric measures.
* Psychiatrist or psychologist to screen for depression, uncontrollable psychosis, suicidal ideation, and hostile or unsupportive family environment.
* Bone age will be obtained to ensure subject has reached or near full growth potential.
* Pediatric Cardiology for echocardiogram to rule out left ventricular hypertrophy.
* Oral glucose tolerance test to assess glucose status and degree of insulin resistance.
* Blood work to assess hepatic and kidney function, nutritional deficiencies, hormonal profile, and hyperlipidemia.
* Pediatric Pulmonary for sleep study and Pulmonary Function Tests (PFTs) to rule out obstructive sleep apnea.

When a subject is approved for surgery, he or she will meet with Bariatric Surgeon to discuss benefits and risks of each bariatric surgery. After the appropriate discussion with surgeon, the choice of procedure will be made by subject and legal guardian. For research purposes, we seek to monitor the progress of the patients enrolled in Yale's Adolescent Bariatric Surgery Clinic. Collecting pre and post long term operative data will allow us to describe this efficacy and potential complications that arise with RYGB vs LAGB.

As standard of care, all subjects will have undergone pre-operative testing established by Adolescent Bariatric Surgery Clinic before any of the bariatric surgeries.

For research purposes:

1. Month prior to Surgery

   * Oral Glucose Tolerance Test (OGTT)
   * Abdominal MRI (weight must not exceed 140 kg)
   * DNA blood extraction

   During RYGB or LAGB Surgery
   * Liver Biopsy
   * Visceral (omental fat) and Subcutaneous Fat Biopsy

   Data collection will continue for 24 months post-operatively and include both research testing and standard of care clinical appointments.

   Post Surgery 2 week 2 months 3 months 6 months 12 months 24 months Standard Of Care Post-op Post-op Post-op Post-op Post-op Post-op Anthropometric X X X X X X Measures Hemoglobin A1c X X X X X
2. Week 2 Month 3 Month 6 Month 12 Month 24 Month Post Surgery (research) Post-op Post-op Post-op Post-op Post-op Post-op OGTT X X X Abdominal MRI X X X X X X

Anthropometric Measures and HBA1c Anthropometric measures will be done at study enrollment, monthly leading up to the surgery RYGB or LAGB, and 2 weeks, 2 months, 3 months, 6 months, 12 months and 24 months post operatively. These measures include height, weight, BMI, BMI Z score, systolic and diastolic blood pressure, resting heart rate, % fat mass, and total fat mass. Demographic data includes ethnicity and family income. HbA1c will be completed at the 3, 6 , 12, and 24 month post operative time period.

ELIGIBILITY:
Inclusion Criteria:

Youth 14-19yrs

* 6 months of attempts at weight management by primary care physician or Pediatric Endocrinologist
* Approval by the Adolescent Bariatric Surgery clinic to undergo surgery
* Physically or nearly physically mature
* BMI >= 35kg/m2 with one obesity related comorbidities or BMI >= 40 kg/m2
* Commitment to avoid pregnancy for at least 1 year postoperatively
* Capability and willingness to adhere to nutritional guidelines postoperatively
* Informed consent to surgical treatment
* Demonstration of decisional capacity
* Supportive family environment

Exclusion Criteria:

* Inability to be approved by Yale Adolescent Bariatric Surgery clinic to undergo surgery
* Uncontrolled psychosis
* Uncontrolled depression
* Drug or alcohol abuse
* History of congenital or acquired anomalies of gastrointestinal tract
* Esophageal anatomical abnormality or dysmotility
* Inflammatory bowel disease
* Severe cardiopulmonary disease
* Severe coagulopathy
* Hepatic insufficiency or cirrhosis
* Presence of localized or systemic infection at time of surgery
* Obesity related to central causes: Prader Willi and hypothalamic abnormalities
* Non-compliance to nutrition plan, exercise, and behavioral counseling/treatment
* Pregnant, breast-feeding or planning of becoming pregnant within 1-2 years of surgery

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The research subjects will be recruited from the Yale Pediatric Obesity Clinic and the Endocrine Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Glucose Tolerance | baseline, 2 month, 3 month, 12 month
  Glucose tolerance changes measured by 3 hour oral glucose tolerance test.

SECONDARY OUTCOMES:
Change in Anthropometric data | Baseline, 2 weeks, 2 mnths, 3 months, 6 months, 12 months, 24 months
  Height, weight, body fat percentage changes
Changes in nutritional health | Baseline, 2 weeks, 2 mnths, 3 months, 6 months, 12 months, 24 months
  Changes in vitamin/mineral blood levels

OTHER OUTCOMES:
Fat distribution | baseline, 2 weeks, 2 months, 3 months, 6 months, 12 months, 24 months
  Abdominal MRI

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale University
Locations (1):
- Yale Pediatric Endocrinology Clinic, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No